CLINICAL TRIAL: NCT05266768
Title: An Open, Single-arm Clinical Study Evaluating the Safety and Efficacy of IBI346 Infusion in Relapsed/Refractory Multiple Myeloma
Brief Title: Study to Evaluate the Safety, Tolerance, Pharmacokinetics and Preliminary Efficacy of IBI346#CIBI346Y002#
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chunrui Li (Other)
Collaborators: Innovent Biologics (Suzhou) Co. Ltd. (Industry)
Responsible Party: Sponsor-Investigator, Chunrui Li, Professor, Tongji Hospital
Organization: Tongji Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIBI346Y002
Record Dates: First submitted 2022-02-23; First posted 2022-03-04 (Actual); Last update posted 2022-11-30 (Actual); Status verified 2022-03

CONDITIONS: Relapsed/Refractory Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- IBI346 (Experimental): Single arm
  Interventions: Drug: IBI346

INTERVENTIONS:
Drug: IBI346 — IBI346 Antibody and IBI346 CAR-T cell injection

SUMMARY:
An open label, single-arm clinical study evaluating the safety and efficacy of IBI346 infusion in relapsed/refractory multiple myeloma

ELIGIBILITY:
Inclusion Criteria:

1. According to the multiple myeloma diagnostic criteria of the International Myeloma Working Group (IMWG), there is the initial diagnosis of multiple myeloma.
2. Subjects must have previously received at least 3 anti-myeloma regimens. Subjects must have documented disease progression (according to IMWG criteria) during or within 12 months of completing their last anti-myeloma regimen prior to study entry; and prior regimens must have included proteasome inhibitor (PI) and immunomodulatory drug (IMiD).
3. Measurable disease as defined by the protocol
4. ECOG score is 0 or 1.
5. Expected survival time ≥12 weeks.

Exclusion Criteria:

1. Patients suffering from graft-versus-host disease (GVHD) or requiring immunosuppressants drugs.
2. Patients who received autologous hematopoietic stem cell transplantation (ASCT) or prior allogeneic hematopoietic stem cell transplantation (ALLo-HSCT) within 12 weeks prior to mononuclear cell collection.
3. No unmobilized mononuclear cells can be collected for CAR T cell production.
4. Screening subjects who were receiving systemic steroids during the previous 7 days or who were determined by the investigator to require long-term systemic steroid use during treatment (except for inhaled or topical use, except at doses < 10mg/ day).
5. Patients with a history of hypertension that cannot be controlled by medication (blood pressure ≥140/90 mmHg).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2022-04-28 (Actual); Primary Completion 2024-02-28 (Estimated); Study Completion 2024-02-28 (Estimated)

PRIMARY OUTCOMES:
Dose limiting toxicity (DLT) | 21 days post IBI346 administration
Incidence and severity of adverse events: Proportion of subjects with treatment-related adverse events assessed by NCI-CTCAE v5.0 criteria | 2 years post IBI346 administration
Presence or absence of replication-competent lentivirus (RCL) | Baseline up to 15 years

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | 3 months post IBI346 administration
  Number of patients with a best response of either complete response, stringent complete response, very good partial response or partial response, assessed using modified International Myeloma Working Group response criteria（2016）
Duration of Response (DOR) | 2 years post IBI346 administration
  DOR will be calculated among responders (with a PR or better response) from the date of initial response (PR or better) to the date of first documented evidence of progressive disease, as defined in the IMWG criteria (2016).
Progression-free Survival (PFS) | 2 years post IBI346 administration
  PFS defined as time from date of initial administration of IBI346 to date of first disease progression according to IMWG criteria (2016), or death due to any cause, whichever occurs first.
Overall Survival (OS) | 2 years post IBI346 administration
  OS is measured from the date of the initial administration of IBI346 to the date of the subject's death.
Pharmacokinetics parameters of IBI346 cells -Maximum CAR level in blood (Cmax) | 2 years post IBI346 administration
Pharmacokinetics parameters of IBI346 cells -Time to peak CAR level in blood (Tmax) | 2 years post IBI346 administration
Pharmacokinetics parameters of IBI346 cells - Area under the curve of the CAR level in blood (AUC) | 2 years post IBI346 administration
Pharmacokinetics parameters of IBI346 antibody- Peak Plasma Concentration (Cmax) | 2 years post IBI346 administration
Pharmacokinetics parameters of IBI346 antibody- Area under the plasma concentration versus time curve (AUC) | 2 years post IBI346 administration
Pharmacokinetics parameters of IBI346 antibody- clearance (CL) | 2 years post IBI346 administration
Pharmacokinetics parameters of IBI346 antibody- half-life (t1/2) | 2 years post IBI346 administration
Pharmacodynamics characteristics - Cytokines Concentrations, cytokines level and the content of soluble BCMA in blood | 2 years post IBI346 administration

CONTACTS AND LOCATIONS:
Overall Officials: Chunrui Li, Principal Investigator — Tongji Hospital
Locations (1):
- Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No